CLINICAL TRIAL: NCT00675805
Title: Prospective Assessment of 0.2 um Pore-sized Filters in Preventing Intravenous Immunoglobulin-associated Adverse Reactions
Brief Title: Preventing Intravenous Immunoglobulin-associated Adverse Reactions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IVIG-001
Record Dates: First submitted 2008-05-07; First posted 2008-05-12 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Immunoglobulin Therapy
Keywords: intravenous immunoglobulin; IVIG; adverse reactions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I (Active Comparator): IVIG infusion with filter
  Interventions: Device: Infusomat filter (Codan Duofilter-Set V86-P)
- Group II (Placebo Comparator): IVIG infusion without filter
  Interventions: Device: IVIG application without filter (Placebo)

INTERVENTIONS:
Device: Infusomat filter (Codan Duofilter-Set V86-P) — An approved filter system may be efficient in retaining complement activating IgG aggregates in IVIG preparations. This effect may reduce complement activation and consecutive inflammation thereby diminishing adverse events during application of intravenous immunoglobulins.
  Other Names: Codan Duofilter-Set V86-P (Ref. 43.4459)
  Arms: Group I
Device: IVIG application without filter (Placebo) — Application Intravenous immunoglobulins without filter (Placebo)
  Arms: Group II

SUMMARY:
In patients treated with the monoclonal antibody infliximab (Remicade®) -which binds to and blocks tumor necrosis factor alpha (TNF-alpha) - an infusomat filter is routinely used to prevent the very same early adverse events observed in individuals receiving intravenous immunoglobulins (IVIG). We recently used such a filter in a patient suffering from malaise and vomiting in the context of an IVIG substitution therapy. In this patient symptoms improved and IVIG-induced complement-activation was reduced (unpublished observation).

Based on this simple observation we hypothesize that this simple and approved filter-system may be efficient in retaining complement-activating immunoglobulin G (IgG) aggregates in IVIG-preparations. This effect may reduce complement activation - and consecutive inflammation - thereby diminishing adverse events.

In this prospective study we propose to investigate how complement activation and side effects after IVIG infusion relate in individuals receiving conventional (i.e. unfiltered) vs. filtered IVIG-preparations.

DETAILED DESCRIPTION:
Prospective single center study with an observational phase (phase A) and a randomized intervention-phase (phase B), monitoring adverse events and complement activation after IVIG infusion. Patients would be enrolled at the Out-patient Clinic of the Division of Hematology at the Department of Internal Medicine at the University Hospital Basel (USB). Based on the number of patients receiving IVIG at the Division of Hematology of the USB we expect to be able to complete data accrual within 8-10 months.

Inclusion criteria: all patients at the Division of Hematology at the University Hospital of Basel, Switzerland after allogeneic stem cell transplant and older than 18 years which are planed for at least 2 applications of IVIG. The patients are included in this study only by informed consent.

Methods: Side effects of IVIG will be monitored by use of a standardized questionnaire distributed to the nursing staff and the patients (please see attachment). Complement activation will be monitored before and after the IVIG-infusion using standard C3, C4 and 50% complement hemolytic activity (CH50) assays. Serum levels of immunoglobulin A, immunoglobulin M and immunoglobulin G will be quantified before and after IVIG-infusion. In phase A of the study we aim at including approximately 40 patients (which would be predicted to include approximately 20 patients with clinical symptoms). In phase B we would randomize these same patients into two groups of similar sizes, the first group receiving standard unfiltered IVIG infusions, the second group receiving 0.2um filtered IVIG infusions

ELIGIBILITY:
Inclusion Criteria:

* All patients at the Division of Hematology at the University Hospital of Basel, Switzerland after allogeneic stem cell transplant and older than 18 years which are planned for at least 2 applications of IVIG. The patients are included in this study only by informed consent.

Exclusion criteria:

* if inclusion criteria not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Measure activity of complement prior to and after completion of IVIG infusion with/without filter (intervention group/placebo group) in these same patients | Prior to and after completion of IVIG infusion with/without filter

SECONDARY OUTCOMES:
Monitor adverse reactions experienced by patients receiving IVIG by use of a standardized questionary | During IVIG infusion

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hess, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Switzerland, Basel, Canton Basel-Town, Switzerland

REFERENCES:
- [Background] Katz U, Achiron A, Sherer Y, Shoenfeld Y. Safety of intravenous immunoglobulin (IVIG) therapy. Autoimmun Rev. 2007 Mar;6(4):257-9. doi: 10.1016/j.autrev.2006.08.011. Epub 2006 Aug 28. PMID 17317619
- [Background] Jarius S, Eichhorn P, Albert MH, Wagenpfeil S, Wick M, Belohradsky BH, Hohlfeld R, Jenne DE, Voltz R. Intravenous immunoglobulins contain naturally occurring antibodies that mimic antineutrophil cytoplasmic antibodies and activate neutrophils in a TNFalpha-dependent and Fc-receptor-independent way. Blood. 2007 May 15;109(10):4376-82. doi: 10.1182/blood-2005-12-019604. Epub 2007 Jan 30. PMID 17264299